CLINICAL TRIAL: NCT06002139
Title: Does Immersive Virtual Reality Therapy Support Orthopedic Rehabilitation? A Randomized-Controlled Trial
Brief Title: Virtual Reality in Orthopedic Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joanna Szczepańska-Gieracha (Other)
Collaborators: Wroclaw Medical University (Other); Wroclaw University of Health and Sport Sciences (Other); Jan Dlugosz University in Czestochowa (Other)
Responsible Party: Sponsor-Investigator, Joanna Szczepańska-Gieracha, Professor, Wroclaw University of Health and Sport Sciences
Organization: Wroclaw University of Health and Sport Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VRortoTrzebnica
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Arthropathy; Anxiety; Stress
Keywords: arthroplasty; stress; fall risk; depression; anxiety; self-efficacy
MeSH Terms: conditions — Joint Diseases; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive Virtual Reality Therapy (Experimental): Conventional orthopedic rehabilitation supplemented by VR therapy
  Interventions: Behavioral: Immersive Virtual Reality Therapy; Behavioral: Conventional rehabilitation
- Conventional rehabilitation (Active Comparator): Conventional orthopedic rehabilitation
  Interventions: Behavioral: Conventional rehabilitation

INTERVENTIONS:
Behavioral: Immersive Virtual Reality Therapy — 8 sessions of VR therapy over 4 weeks (each of them 20 minutes long).
  As a virtual reality source, VRTierOne device (Stolgraf®) were used. Thanks to using head mounted display and the phenomenon of total immersion VR therapy provides an intense visual, auditory and kinesthetic stimulation. It can have a calming and mood-improving effect or help the patients recognize their psychological resources and motivate to the rehabilitation process. In the virtual therapeutic garden there are a rich set of symbols and metaphors based on Ericksonian Psychotherapy approach. The most important is the Garden of Revival which symbolizes the patient's health. It used to be full of life and energy, now it is neglected, requires work to be revived. In the therapeutic process day by day, the therapist tells the patient a symbolic story about his/her situation.
  Arms: Immersive Virtual Reality Therapy
Behavioral: Conventional rehabilitation — Four weeks of conventional rehabilitation including:
  * Two hours of kinesiotherapy (120 minutes, including gait training).
  * Thirty minutes of ergotherapy.
  * Three physical therapy procedures (i.e. laser therapy, magnetic therapy, electrotherapy) tailored to individual ailments and needs.

SUMMARY:
The study's objective is to evaluate the efficacy of implemented Virtual Reality therapy for patients who have undergone lower limb arthroplasty and are in inpatient rehabilitation. The study aim to examine its influence on reducing anxiety levels, mitigating depressive symptoms, enhancing motivation for elderly patients to participate in physiotherapy, and improving their overall functional state and fall risk.

DETAILED DESCRIPTION:
The study will include elderly patients (60+) who present sequentially at the General Systemic Rehabilitation Department of St. Hedwig of Silesia Hospital in Trzebnica, within 3 months of having undergone hip or knee joint arthroplasty surgery. Patients will be randomly assigned to one of two groups: A. Virtual Reality Group: 8 therapy sessions, two sessions per week; B. Control group, undergoing conventional rehabilitation. Participation in the study is entirely voluntary, and written consent is required.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have recently undergone hip or knee joint arthroplasty surgeries aged 60 years and above.

Exclusion Criteria:

* cognitive impairments that prevent independent completion of research questionnaires
* reported consciousness disorders
* bipolar affective disorder and other serious mental disorders in the patient's medical history
* use of psychoactive drugs
* ongoing psychiatric treatment or individual psychological therapy
* contraindications to Virtual Reality such as epilepsy, vertigo, serious vision disorders
* functional status preventing independent movement (orthopedic aids are allowed, e.g., crutches, walker)
* refusal to participate in the study at any stage

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | 15 minutes
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale scoring from 0 to 3 for each item. The first seven items relate to anxiety (HADS-A), and the remaining seven items relate to depression (HADS-D). The global scoring ranges from 0 to 42 with a cut-off point of 8/21 for anxiety and 8/21 for depression. The higher the score, the greater anxiety or depression symptoms.
Perceived Stress Scale | 10 minutes
  The Perceived Stress Scale (PSS-10) is a ten-item scale that assesses the level of stress perceived by an individual in the last month. The questions are general in nature and fairly free of content specific to any subpopulation group. The items are designed to tap into how unpredictable, uncontrollable, and overloaded respondents find their lives to be. The scores range from 0 to 40, with higher scores indicating higher perceived stress. The Perceived Stress Scale will be administered at the beginning and after four weeks of treatment.

SECONDARY OUTCOMES:
Generalized Self-Efficacy Scale | 15 minutes
  The Generalized Self-Efficacy Scale (GSES) is a ten-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. The scale measures the belief in one's competence to cope with a broad range of stressful or challenging demands. The score ranges from 10 to 40, with a higher score indicating a greater sense of self-efficacy. The Generalized Self-Efficacy Scale will be applied at the beginning and after four weeks of treatment.
Barthel Index | 15 minutes
  The Barthel Index (BI) is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. It uses ten variables describing activities of daily living and mobility. Scores range from 0 to 100, with higher scores associated with a greater likelihood of being able to live at home with a degree of independence following discharge from the hospital. The the Barthel Index will be administered at the beginning and after four weeks of treatment.
Rivermead Mobility Index | 15 minutes
  The Rivermead Mobility Index (RMI) was developed from the Rivermead Motor Assessment Gross Function subscale as a means to quantify mobility disability. It is composed of 14 items representing different mobility tasks, ranging from turning over in bed to running. Each item is scored as 'unable' (0) or 'able' (1), leading to a maximum score of 14, which indicates full mobility. The Rivermead Mobility Index will be administered at the beginning and after four weeks of treatment.
Tinetti's Short Scale | 15 minutes
  Tinetti's Short Scale for fall risk assessment is a shortened version of Performance-Oriented Mobility Assessment (POMA). It is easily administered test that measures a patient's gait and balance. The test is scored on the patient's ability to perform following tasks: Change from sitting to standing, Immobilization in standing position for 5 seconds, Passing 3 meters, Turn of 180 degrees, Keeping a sitting position. Each task is rated in 3-point Likert scale. The scales rage from 0-15, with the higher scores indicate better functional mobility.
Short Physical Performance Battery | 15 minutes
  The Short Physical Performance Battery (SPPB) is a group of measures that combines the results of the gait speed, chair stand and balance tests. It provides a composite score ranging from 0 (worst performance) to 12 (best performance), offering a global assessment of physical functioning in older individuals. The SPPB will be administered at the beginning and after four weeks of treatment.
Perception of Stress Questionnaire | 20 minutes
  The Perception of Stress Questionnaire (PSQ) was created by Plopa and Makarowski. It is a 27-item scale scoring from 1 to 5 points for each item, where 21 items examine the level of stress in the areas of emotional tension, external stress and intrapsychic stress, and six items refer to the lie scale. The global scoring for the perception of stress ranges from 21 to 105, with a cut-off point of 60 for an elevated level of perceived stress. Higher scores indicate higher stress perception.

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Mazurek, PhD, Study Chair — Wroclaw Medical University; Błażej Cieślik, PhD, Study Chair — Jan Dlugosz University in Czestochowa, Poland; Justyna Mazurek, RhD, Principal Investigator — Wroclaw Medical University; Joanna Szczepańska-Gieracha, Professor, Study Director — Wrocław University of Health and Sport Sciences; Robert Gajda, PhD, Study Director — Gajda-Med District Hospital in Pułtusk
Locations (1):
- St. Hedwig of Silesia Hospital in Trzebnica, Trzebnica, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cieslik B, Mazurek J, Rutkowski S, Kiper P, Turolla A, Szczepanska-Gieracha J. Virtual reality in psychiatric disorders: A systematic review of reviews. Complement Ther Med. 2020 Aug;52:102480. doi: 10.1016/j.ctim.2020.102480. Epub 2020 Jun 9. PMID 32951730
- [Background] Rutkowski S, Kiper P, Cacciante L, Cieslik B, Mazurek J, Turolla A, Szczepanska-Gieracha J. Use of virtual reality-based training in different fields of rehabilitation: A systematic review and meta-analysis. J Rehabil Med. 2020 Nov 19;52(11):jrm00121. doi: 10.2340/16501977-2755. PMID 33073855
- [Background] Kiper P, Przysiezna E, Cieslik B, Broniec-Siekaniec K, Kucinska A, Szczygiel J, Turek K, Gajda R, Szczepanska-Gieracha J. Effects of Immersive Virtual Therapy as a Method Supporting Recovery of Depressive Symptoms in Post-Stroke Rehabilitation: Randomized Controlled Trial. Clin Interv Aging. 2022 Nov 23;17:1673-1685. doi: 10.2147/CIA.S375754. eCollection 2022. PMID 36447623
- [Background] Szczepanska-Gieracha J, Cieslik B, Rutkowski S, Kiper P, Turolla A. What can virtual reality offer to stroke patients? A narrative review of the literature. NeuroRehabilitation. 2020;47(2):109-120. doi: 10.3233/NRE-203209. PMID 32741792
- [Background] Czech O, Siewierska K, Krzywinska A, Skorniak J, Maciejczyk A, Matkowski R, Szczepanska-Gieracha J, Malicka I. Virtual Therapy Complementary Prehabilitation of Women Diagnosed with Breast Cancer-A Pilot Study. Int J Environ Res Public Health. 2022 Dec 30;20(1):722. doi: 10.3390/ijerph20010722. PMID 36613047
- [Background] Szczepanska-Gieracha J, Jozwik S, Cieslik B, Mazurek J, Gajda R. Immersive Virtual Reality Therapy as a Support for Cardiac Rehabilitation: A Pilot Randomized-Controlled Trial. Cyberpsychol Behav Soc Netw. 2021 Aug;24(8):543-549. doi: 10.1089/cyber.2020.0297. Epub 2021 Feb 11. PMID 33577375
- [Background] Cieslik B, Juszko K, Kiper P, Szczepanska-Gieracha J. Immersive virtual reality as support for the mental health of elderly women: a randomized controlled trial. Virtual Real. 2023 May 7:1-9. doi: 10.1007/s10055-023-00797-w. Online ahead of print. PMID 37360811
- [Background] Rutkowski S, Szczegielniak J, Szczepanska-Gieracha J. Evaluation of the Efficacy of Immersive Virtual Reality Therapy as a Method Supporting Pulmonary Rehabilitation: A Randomized Controlled Trial. J Clin Med. 2021 Jan 18;10(2):352. doi: 10.3390/jcm10020352. PMID 33477733